CLINICAL TRIAL: NCT03452800
Title: Work on the Social Representation of Addiction Among Mental Health Professionals
Brief Title: Addiction Among Mental Health Professionals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7014
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-02

CONDITIONS: Addiction
Keywords: addiction; mental health
MeSH Terms: conditions — Behavior, Addictive; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our goal is to determine the representations of addiction among caregivers working in the field of mental health. We hypothesize that caregivers, despite their investment in care, have a negative social representation of patients suffering from addictive disorders, which could be related to a lack of training on the pathology and its social repercussions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Health professional with more than 5 years of professional experience in the field of management of mental illnesses
* Health professional having accepted to participate in the study

Exclusion Criteria:

- Refusal to participate in the stud

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health professional with more than 5 years of professional experience in the field of management of mental illnesses
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Number of addictions | Period from 5 years of professional experience will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LALANNE-TONGIO, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Psychiatrie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No